CLINICAL TRIAL: NCT04310137
Title: The Effect of Self-directed Versus Therapist-directed Re-loading on Incidence of Ulcer Recurrence
Brief Title: Self-directed Versus Therapist-directed Re-loading on Incidence of Ulcer Recurrence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercer University (Other)
Responsible Party: Principal Investigator, Deborah M. Wendland, Ph.D., Associate Professor, Mercer University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H1908191
Record Dates: First submitted 2020-02-19; First posted 2020-03-17 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; re-loading; ulcer recurrence
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be unaware of in which group the participant was randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapist-Directed Re-loading (Experimental): Participants in this arm will be instructed to increase their activity by walking 10% more steps per day than the steps recorded in the most recent activity monitoring (i.e. StepWatch) measurement (e.g. 10% more than the initial monitoring values and 10% more than the second monitoring values once they are completed).
  Interventions: Behavioral: Therapist-Directed Re-loading
- Self-Directed Re-loading (No Intervention): Participants in this arm will be instructed to slowly increase their walking.

INTERVENTIONS:
Behavioral: Therapist-Directed Re-loading — Therapist will specifically direct participant to increase walking by 10% as measured at each of the activity monitoring assessments. In addition, the participant will be asked to monitor foot temperature to mitigate risk for breakdown.
  Arms: Therapist-Directed Re-loading

SUMMARY:
This study is designed to evaluate if how people are told to return to walking after a skin injury affects whether or not they develop new (recurrence) skin breakdown on their feet. The people in this study will have diabetes and have a recently closed foot ulcer. About half will be specifically told how to return to walking and the other half will be told to return to walking slowly. How people naturally return to walking will also be established.

DETAILED DESCRIPTION:
The purpose of this project is to determine the impact of Therapist-directed loading versus self-selected loading on ulcer occurrence and to establish natural loading behavior following diabetic foot ulcer closure.

Eligible participants will be randomized into a group given specific directions from a Therapist to return to walking (i.e. reloading skin following plantar ulceration closure) or a group encouraged to slowly return to walking (self-directed re-loading of the skin following plantar ulceration closure). Following randomization and instruction for re-loading according to group assignment, participants will be assessed every 6 months for walking behavior. Participants will be monitored for ulcer recurrence throughout. Participants will be followed for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* With or without peripheral neuropathy
* Able to safely exercise
* Have a recently closed plantar ulceration

Exclusion Criteria:

* Presence of an open plantar ulceration
* Presence of an untreated infection
* Presence of osteomyelitis or gangrene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ulcer Recurrence | Over up to 18 months of follow-up.
  Assessment of incidence of any plantarr ulcer recurrence.
Change in walking behavior (steps) | Assessed initially and every 6 months for 1 week for up to 18 months.
  Actual assessment of change in walking behavior will be assessed by number of steps.
Change in walking behavior (step timing) | Assessed initially and every 6 months for 1 week for up to 18 months.
  Actual assessment of change in walking behavior will be assessed by the timing of steps (how many steps in a given timeframe).

SECONDARY OUTCOMES:
Exercise component of Summary of Diabetes Self-Care Activities Scale | Assessed initially and every 6 months for up to 18 months
  Questionnaire to assess exercise adherence. It is a report of the number of days that an individual participates in physical activity as well as specific exercise (2 questions). The higher the number, the more days of activity/exercise participation. The more days of participation, the better the investigators would expect health to be.
Bio-thesiometer | Assessed initially and every 6 months for up to 18 months
  Assesses vibration sense
Body Mass Index (BMI) and disease risk | Assessed initially and every 6 months for up to 18 months
  Weight and height will be combined to report BMI in kg/m^2.
Waist circumference | Assessed initially and every 6 months for up to 18 months
  Waist circumference (measured in cm) will be assessed for change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M. Wendland, Principal Investigator — Mercer University
Locations (1):
- Piedmont Healthcare, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified step data will be made available through a repository upon conclusion of the study and its dissemination.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following the study conclusion and its dissemination (6 months after publication).
Access Criteria: This information will be shared with researchers for meta-analyses through the data repository.